CLINICAL TRIAL: NCT01562652
Title: AposTherapy for Singaporean Patients With Knee Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apos_Sing_01
Record Dates: First submitted 2012-03-14; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- Research (Experimental)
  Interventions: Device: AposTherapy (All Phases of Step-cycle {APOS} system, APOS-Medical and Sports Technologies Ltd. Herzliya, Israel)

INTERVENTIONS:
Device: AposTherapy (All Phases of Step-cycle {APOS} system, APOS-Medical and Sports Technologies Ltd. Herzliya, Israel)

SUMMARY:
Osteoarthritis (OA) is the most prevalent form of arthritis in the elderly. It is estimated that 7% of men and 11% of women over the age of 65 have KOA. The most significant symptoms of the disease are pain and functional disability.

This study has two aims:

1. To characterise the gait patterns and clinical parameters of patients with knee osteoarthritis (KOA) in Singapore at baseline, prior to treatment.
2. To investigate the changes in gait patterns and the clinical benefits of treatment with a new biomechanical device, AposTherapy, for patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic bilateral knee osteoarthritis at the medial compartment for at least six months, fulfilling the ACR clinical criteria for OA of the knee, and having radiographically assessed OA of the knee according to the Kellgren and Lawrence scale.
* Patients with an overall WOMAC score of >2cm (as measured at baseline).
* Males and females between the ages of 50-70.

Exclusion Criteria:

* Patients suffering from acute septic arthritis.
* Patients suffering from inflammatory arthritis.
* Patients who received a corticosteroid injection within 3 months of the study.
* Patients suffering from avascular necrosis of the knee.
* Patients with a history of knee buckling or recent knee injury.
* Patients who have had a joint replacement.
* Patients suffering from neuropathic arthropathy.
* Patients with an increased tendency to fall.
* Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedure.
* Patients with a history of pathological osteoporotic fracture.
* Patients suffering from symptomatic degenerative arthritis in lower limb joints other than the knees.
* Patients with referred pain in the knees from back or hip joint symptoms.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)

PRIMARY OUTCOMES:
Changes in self-evaluation questionnaires between baseline and after 6 months of therapy | Baseline, 6 months
  Western Ontario and MacMaster osteoarthritis questionnaire (WOMAC) and SF-36 Health Survey will be evaluated.
  The WOMAC questionnaire is measured on a 10cm visual analogue scale (VAS) and the SF-36 is scored between 0-100.

SECONDARY OUTCOMES:
Changes in spatio-temporal gait parameters between basline and after 6 months of therapy | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Aloni, Principal Investigator — AposTherapy Singapore Pte Ltd. #05-07, 1 Orchard Boulevard Singapore 248649
Locations (1):
- AposTherapy center, Singapore, Singapore

REFERENCES:
- [Derived] Elbaz A, Mor A, Segal G, Aloni Y, Teo YH, Teo YS, Das-De S, Yeo SJ. Patients with knee osteoarthritis demonstrate improved gait pattern and reduced pain following a non-invasive biomechanical therapy: a prospective multi-centre study on Singaporean population. J Orthop Surg Res. 2014 Jan 2;9:1. doi: 10.1186/1749-799X-9-1. PMID 24383821